CLINICAL TRIAL: NCT05208268
Title: A Post-marketing Surveillance of Pariet Tab. 5 mg to Prevent Gastric and Duodenal Ulcer Associated With Low-aspirin, 100 mg or Less Daily, Administration in Korean Patients With a History of Gastric and Duodenal Ulcer
Brief Title: A Study of Pariet to Prevent Gastric and Duodenal Ulcer Associated With Low-aspirin in Korean Participants With a History of Gastric and Duodenal Ulcer
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E3810-M082-520
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-01

CONDITIONS: Stomach Ulcer; Duodenal Ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pariet: Participants with gastric and duodenal ulcer being administered with Pariet 5 mg, tablet within the scope of the approved label for Korea under the medical judgment of the investigator will be observed up to maximum of 24 weeks.
  Interventions: Drug: Pariet

INTERVENTIONS:
Drug: Pariet — Pariet Tablets.
  Other Names: Rabeprazole Sodium

SUMMARY:
The purpose of this study is to understand the following safety related particulars associated with the use of Pariet Tablet 5 milligram (mg) to prevent gastric and duodenal ulcer from low dose aspirin administration of 100 mg or less daily in participants with a history of gastric and duodenal ulcer: 1. Serious adverse events (SAEs) and adverse drug reactions (ADRs) 2. Unexpected adverse events (AEs) and ADRs not reflected in the precautions for use 3. Known ADRs 4. Non-serious ADRs 5. Other safety and efficacy related information.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged over 18 years
2. Participants who have a history of gastric and duodenal ulcer falling under the approved indication for Pariet Tablet 5 mg and who are receiving Pariet Tablet 5 mg to prevent gastric and duodenal ulcer from low dose aspirin use of 100 mg or less daily
3. Participants whose prescription of Pariet Tablet 5 mg has been determined before study participation
4. Participants who have given written consent to the use of their personal and medical information

Exclusion Criteria:

1. Participants with a known hypersensitivity to rabeprazole sodium, any excipients used in the formulation or benzimidazole derivatives, and with the history of such hypersensitivity
2. Participants administered with atazanavir
3. Pregnant or lactating
4. Participants administered with rilpivirine
5. Participants currently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with gastric and duodenal ulcer who have been administered with Pariet 5 mg will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With SAEs | Up to Week 24
  SAEs is defined as any untoward medical occurrence: resulting in death; life threatening condition requiring hospitalization or prolongation of hospitalization; resulting in persistent or significant disability or incapacity; resulting in birth defect or occurrence of other medically significant events that need treatment such as drug dependency or abuse, blood disease.
Percentage of Participants With ADRs | Up to Week 24
  An ADR is defined as all noxious and unintended responses to a study drug related to any dose. All adverse events in which its causal relationship with the study drug is at least a reasonable possibility will be reported as ADR.
Percentage of Participants With Unexpected AEs | Up to Week 24
  An AE is defined as any untoward and unintended signs (example, anomalies in laboratory test results), symptoms, or diseases occurring during administration of drug, which do not necessarily have a causal relationship with the drug in question. An unexpected AE is an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug.
Percentage of Participants With Unexpected ADRs | Up to Week 24
  An ADR is defined as all noxious and unintended responses to a study drug related to any dose. All adverse events in which its causal relationship with the study drug is at least a reasonable possibility will be reported as ADR. An unexpected ADR is an ADR with difference in the nature or severity, specificity, or the outcome, compared to the product licensure/notification of the drug.
Percentage of Participants With Already Known ADRs | Up to Week 24
  An ADR is defined as all noxious and unintended responses to a study drug related to any dose. All adverse events in which its causal relationship with the study drug is at least a reasonable possibility will be reported as ADR. Already known ADRs are those listed in product licensure/notification of the drug.
Percentage of Participants With Non-serious ADRs | Up to Week 24
  An ADR is defined as all noxious and unintended responses to a study drug related to any dose. All adverse events in which its causal relationship with the study drug is at least a reasonable possibility will be reported as ADRs.
Percentage of Participants with Final Effectiveness Evaluation | Up to Week 24
  Participants assessed for final effectiveness after first dose of drug will be categorized into four categories: Improved, Unchanged, Worsened, and Unknown.

CONTACTS AND LOCATIONS:
Locations (29):
- South Korea (29):
  - Site #09, Bucheon-si, Gyeongji-do
  - Site #31, Bucheon-si, Gyeongji-do
  - Site #24, Dongtan, Gyeongji-do
  - Site #03, Ilsan, Gyeongji-do
  - Site #11, Ilsan, Gyeongji-do
  - Site #17, Incheon, Gyeongji-do
  - Site #20, Changwon, Gyeongsangnam-do
  - Site #29, Iksan, Jeollabuk-do
  - Site #19, Cheongju-si, North Chungcheong
  - Site #01, Chungju, North Chungcheong
  - Site #07, Busan
  - Site #08, Busan
  - Site #14, Busan
  - Site #15, Busan
  - Site #28, Busan
  - Site #02, Daegu
  - Site #23, Daegu
  - Site #27, Daegu
  - Site #05, Seoul
  - Site #06, Seoul
  - Site #10, Seoul
  - Site #13, Seoul
  - Site #16, Seoul
  - Site #18, Seoul
  - Site #21, Seoul
  - Site #22, Seoul
  - Site #25, Seoul
  - Site #26, Seoul
  - Site #30, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.